CLINICAL TRIAL: NCT00811278
Title: A Non-Invasive Approach to Predict Steroid Sensitivity in Patients With Asthma
Brief Title: Approach to Predict Steroid Sensitivity in Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 08-50
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: inhaled corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- step1: asthma patients on step 1 therapy
- step 2: asthma patients on step 2 therapy
- healthy: non-asthmatics

SUMMARY:
Inhaled corticosteroids are widely used as the primary therapy for asthma, which affects approximately 20 million people in the United States. While many patients respond to corticosteroid therapy, as many as 25-30% of patients with severe asthma have asthma that is difficult to treat or steroid insensitive. Predictive biomarkers for the rapid identification of patients with asthma who will achieve adequate control of their symptoms with inhaled corticosteroids has the potential to significantly improve asthma management. This proposal is based on the hypothesis that alterations in gene expression in epithelial cells of the buccal mucosa can be used as a reliable biomarker to predict corticosteroid response in patients with asthma. The goals of this proposal will determine if gene expression in epithelial cells of the buccal mucosa from patients with asthma is in concordance with gene expression profiles that have been identified through more invasive sampling techniques of the airway epithelium of asthma patients. The Specific Aims of this proposal are to 1) investigate the level of variability in gene expression of a subset of inflammatory markers in buccal epithelium from adult patients with asthma. Aim 1 will be carried out by collecting buccal samples from three cohorts of subjects (18-55 years of age) from the Pulmonology and Allergy Clinics at Truman Medical Center during regularly scheduled outpatient visits as follows: 1) healthy control adult subjects (n=10), 2) patients with asthma treated only with a short-acting beta2-agonist (SABA, n=10), and 3) patients with asthma treated with low-dose ICS (n=10). Relative gene expression of inflammatory markers will be determined using quantitative RT (reverse transcription)-PCR and variability in gene expression will be determined within and between the three cohorts. Data from the pilot studies described in this proposal will aid in the determination of appropriate study population sizes for future investigations with the long-term objective to use changes in gene expression (in buccal epithelial cells) as a dynamic biomarker for determining corticosteroid response in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. healthy control adult subjects (n=10),
2. patients with mild to moderate asthma (n=20) (Table 2, Appendix 4).

A diagnosis of asthma will be defined as episodic airflow obstruction which is reversible (improvement in FEV1 >12% when measured via spirometry) after administration of a SABA.

Exclusion Criteria:

1. currently smokers or have been smokers in the past 6 months
2. a diagnosis of COPD, bronchiectasis, Allergic Bronchopulmonary Aspergillosis, diagnosis of bacterial, fungal, or viral pneumonia in the past 6 months, or other diagnoses of chronic lung disease.
3. subjects being treated with oral systemic corticosteroids for other diseases, those using intranasal steroids in a 2 week period preceding the study, or those requiring an oral corticosteroid burst in the past 6 weeks, or who are receiving treatment with immune modulator medications will also be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of the allergy and asthma clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Validation of this technique as a reliable marker for inflammatory expression related to asthma and corticosteroid response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette L. Jones, MD, Principal Investigator — Children's Mercy Hospital and Clinics; Carrie Vyhlidal, PhD, Principal Investigator — Children's Mercy Hospital's and Clinics
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States